CLINICAL TRIAL: NCT05098704
Title: Phase II/III Double-blind Randomized Placebo-controlled Trial Assessing the Preventive Effect of Clopidogrel on the Systemic Sclerosis Development Risk in Subjects With Specific Dysimmunity and Raynaud Phenomenon
Brief Title: Preventive Effect of Clopidogrel on the Systemic Sclerosis Development Risk
Acronym: PSSIT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry for Health and Solidarity, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHUBX 2017/45
Record Dates: First submitted 2021-10-04; First posted 2021-10-28 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Scleroderma; Systemic Sclerosis
Keywords: systemic sclerosis; clopidogrel; platelet; prevention; primary care
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clopidogrel (Experimental)
  Interventions: Drug: clopidogrel treatment
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: clopidogrel treatment — 75 mg daily during 24 months
  Arms: clopidogrel
Drug: Placebo — 75 mg daily during 24 months
  Arms: placebo

SUMMARY:
Systemic sclerosis (SSc) is a severe autoimmune disease associating dysimmunity, vasculopathy and fibrosis. No curative treatment is available. Pre-clinical abnormalities can be found such as specific autoantibodies. The association of Raynaud phenomenon and SSc-specific anti-nuclear antibodies is the hallmark of pre-scleroderma subjects, among who around 47% declare a complete disease after five years. The aim of this study is to assess in this particular population the preventive effect of an anti-platelet treatment.

DETAILED DESCRIPTION:
In this study, platelet activation is targeted as it could play a key role in the pathogenesis of SSc. It has been shown in several publications that platelets are activated in SSc with a correlation between the level of activation and disease activity. Secondary to this activation, soluble and membrane effectors were increased, and induced vascular damages and fibrosis. The results obtained in the laboratory (CNRS UMR-5164) directly involved platelets in this mechanism by inducing the thymic stromal lymphopoietin (TSLP) production by endothelial cells and by showing the pro-fibrotic effect of TSLP. In vivo data in SSc murine model recently obtained, confirmed the preventive role on fibrosis of clopidogrel. The early control of this platelet activation could prevent the course of events leading to SSc.

The therapeutic strategy assessed in this study will be the oral administration of clopidogrel (75 mg per day) during two years to subjects presenting an association of specific dysimmunity and Raynaud phenomenon (RP). The administration of clopidogrel will be double-blinded versus placebo.

Subjects will be included and treated during a 2-year period and will be followed for a period of 36 months after treatment, i.e. a total of 60 months. The follow-up will be every six months mainly comprising clinical examination, patient reported outcomes and blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old, and less than 85 years old.
* Patient with positive AAN (AAN ≥ 1/160) with the following specificity: anti-Scl70 or anti-centromere or anti-RNApolIII, or any other auto-antibodies related to systemic sclerosis
* Patient with RP reported by the subject and confirmed by the physician.
* Patient affiliated to a health insurance system.
* Patient who accepts to participate to the study and signs an inform consent form.

Exclusion Criteria:

* Patient with an SSc diagnosis according to ACR/EULAR 2013 criteria.
* Patient with skin fibrosis at screening.
* Patient with antiplatelet treatment at screening.
* Patient with contraindications to clopidogrel.
* Patient treated by immunosuppressive agent at screening.
* Patient treated by anticoagulants at screening
* Pregnant or breastfeeding women.
* Women of childbearing age refusing effective contraception method during the study treatment (24 months).
* Incompetent adults (i.e. Individuals under the protection of a conservator)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2031-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of occurrence of SSc at 5 years according to American College of Rheumatology (ACR) / European League Against Rhumatism (EULAR) 2013 criteria in the two randomization groups | 60 months after baseline (Day 0)

SECONDARY OUTCOMES:
Frequency of occurrence of cutaneous fibrosis (sclerodactyly or other affected area) clinically assessed by at least 2 independent investigators in the two randomization groups | 60 months after baseline (Day 0)
Mean of modified Rodnan skin score (which varies between 0 and 51, with higher values mean higher disease severity) in the two randomization groups. | 60 months after baseline (Day 0)
Mean of Cochin hand function scale (which varies between 0 and 90, with higher values mean higher disease severity) in the two randomization groups. | 60 months after baseline (Day 0)
Proportion of sex ratio at inclusion in the two randomization groups. | At baseline (Day 0)
Mean age at inclusion in the two randomization groups. | At baseline (Day 0)
Proportion of patients exposed to toxic products at inclusion in the two randomization groups. | At baseline (Day 0)
Proportion of patients exposed to toxic products at 5 years in the two randomization groups. | 60 months after baseline (Day 0)
Proportion of patients affected by a limited form of SSc at 5 years in the two randomization groups. | 60 months after baseline (Day 0)
Proportion of patients affected by a diffuse form of SSc at 5 years in the two randomization groups. | 60 months after baseline (Day 0)
Proportion of patients presenting a specific antibody positivity (anti-scl70, anti-centromere) in the two randomization groups at inclusion. | At baseline (Day 0)
Proportion of patients presenting megacapillaries by capillaroscopy at 5 years in the two randomization groups. | 60 months after baseline (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Elise TRUCHETET, Prof, Principal Investigator — University Hospital, Bordeaux; Linda WITTKOP, MD, Study Chair — University of Bordeaux
Locations (10):
- France (10):
  - CH de la Cote Basque - service de rhumatologie, Bayonne
  - CHU de Bordeaux - service de Médecine Interne et Maladies Infectieuses, Bordeaux
  - CHU de Bordeaux - service de rhumatologie, Bordeaux
  - CHU de Brest - service de rhumatologie, Brest
  - CHU de Grenoble Alpes - service de médecine vasculaire, Grenoble
  - CH de Libourne - service de rhumatologie, Libourne
  - CH de Mont-de-Marsan - service de rhumatologie, Mont-de-Marsan
  - AP-HP - Hôpital Cochin - service de médecine interne, Paris
  - CH de Pau - service de médecine interne, Pau
  - CHU de Toulouse - service de médecine interne, Toulouse